CLINICAL TRIAL: NCT06269094
Title: A Consumer Pilot Study to Understand How Continuous Glucose Monitors Impact Eating Behavior in Individuals Attempting to Lose Weight
Brief Title: A Study to Understand How Continuous Glucose Monitors Impact Eating Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MB-2312
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGM (Experimental)
  Interventions: Other: CGM

INTERVENTIONS:
Other: CGM — CGM use for 6 weeks during virtual focus groups

SUMMARY:
The purpose of this study is to evaluate if and how continuous glucose monitors (CGMs) impact food consumption, choice, and purchasing in individuals attempting to lose weight using their own weight management approach.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-60 y of age.
2. Individual is attempting to lose ≥15 lbs.
3. Individual is able to articulate a weight loss plan.
4. Individual is a primary or co-primary grocery shopper (i.e., does all or most of the grocery shopping for the household or shares the responsibility with someone else).
5. Individual shops for household food and beverages at mainstream grocery stores (e.g., Walmart, Target, Publix, Aldi, Costco, Sam's Club, etc.).
6. Individual consumes packaged food within ≥2 General Mills categories (cereal, bars, yogurt, and soups).
7. Individual has attained a high school diploma or a General Educational Development (GED) equivalent.
8. Individual has a household income ≥$30,000 per year before taxes.
9. Individual has not participated in another research study within 1 month of the screening visit.
10. Individual has access to reliable technology and high-speed internet to attend virtual focus groups and review CGM data in real-time.
11. Individual is willing and able to undergo the scheduled study procedures, including use of a CGM for 6 weeks, complete food logs, answer weekly survey questions, and participate in online group discussions.
12. Individual understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Individual or someone in the household works as a registered dietitian or fitness professional.
2. Individual or someone in the household works for a medical device company for diabetes management.
3. Individual or someone in the household works in the medical field as a nurse, medical doctor, physician assistant, or a close equivalent.
4. Individual or someone in the household currently uses a CGM.
5. Individual has a clinically significant endocrine (e.g., diabetes) or gastrointestinal condition that could interfere with the interpretation of the study results.
6. Individual has a history of cancer in the prior 2 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
7. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening.
8. Individual has a history of a diagnosed eating disorder (e.g., anorexia or bulimia nervosa).
9. Individual has a history of bariatric surgery.
10. Individual is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
11. Individual has a current or recent history (past 12 months of screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
12. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Qualitative insights on consumer behavior | 6 weeks
  Discussions during the virtual focus groups will provide qualitative insights on if/how consumer behavior (related to food choice, eating behavior, and purchasing) changes when using a CGM.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — MB Clinical Research and Consulting LLC
Locations (1):
- Biofortis, Inc., Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No